CLINICAL TRIAL: NCT05501717
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study of Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Subcutaneous ALXN2030 in Healthy Participants
Brief Title: Safety, PK/PD, and Immunogenicity Study of SC ALXN2030 in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALXN2030-HV-101
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ALXN2030 Dose A (Experimental): ALXN2030 will be administered as a single dose.
  Interventions: Drug: ALXN2030
- ALXN2030 Dose B (Experimental): ALXN2030 will be administered as a single dose.
  Interventions: Drug: ALXN2030
- ALXN2030 Dose C (Experimental): ALXN2030 will be administered as a single dose.
  Interventions: Drug: ALXN2030
- ALXN2030 Dose D (Experimental): ALXN2030 will be administered as a single dose.
  Interventions: Drug: ALXN2030
- ALXN2030 Dose E (Experimental): ALXN2030 will be administered as a single dose.
  Interventions: Drug: ALXN2030
- Placebo (Placebo Comparator): Placebo will be administered as a single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN2030 — ALXN2030 will be administered subcutaneously as a single dose either as a manual SC injection or as an SC infusion via a syringe pump.
  Arms: ALXN2030 Dose A; ALXN2030 Dose B; ALXN2030 Dose C; ALXN2030 Dose D; ALXN2030 Dose E
Drug: Placebo — Placebo will be administered subcutaneously as a single dose either as a manual SC injection or as an SC infusion via a syringe pump.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of single ascending doses of ALXN2030 in healthy participants.

DETAILED DESCRIPTION:
Approximately 48 healthy adult participants (36 participants will be on ALXN2030 and 12 participants will be on placebo) are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* QTcF ≤ 450 msec at Screening and on admission (ie, on Day -1).
* Participants of Japanese descent are defined as: First generation (born to 2 Japanese parents and 4 Japanese grandparents).
* Participants of Japanese descent must be between 20 and 60 years of age.
* BMI within the range 18-32kg/m2 (inclusive) at Screening.

Exclusion Criteria:

* Current or recurrent disease
* Current or relevant history of physical or psychiatric illness.
* Any other significant disease or disorder that, in the opinion of the Investigator, may put the participant at risk.
* Female participants who are pregnant or breastfeeding.
* Major surgery or hospitalization within 90 days prior to dosing on Day1.
* History of allergy or hypersensitivity to an oligonucleotide or GalNAc moiety or any excipients of ALXN2030.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | Day 1 through through study completion, an average of 1 year

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Days 1 (predose; end of infusion (EOI); and 0.25, 0.5, 1, 2, 4, 6, 8, and 12 hours post-EOI), 2, 3, 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, and 127
Time to Maximum Observed Plasma Concentration (Tmax) | Days 1 (predose; EOI; and 0.25, 0.5, 1, 2, 4, 6, 8, and 12 hours post-EOI), 2, 3, 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, and 127
Area Under the Plasma Concentration Versus Time Curve From Time 0 (Dosing) to the Last Quantifiable Concentration (AUCt) | Days 1 (predose; EOI; and 0.25, 0.5, 1, 2, 4, 6, 8, and 12 hours post-EOI), 2, 3, 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, and 127
Change from Baseline in Plasma Concentration of Complement Component 3 (C3) Protein | Baseline (Day 1) and study completion, an average of 1 year
Change from Baseline in Serum Complement Functional Activity | Baseline (Day 1) and Day 127
Number of Participants With Treatment-Emergent Antidrug Antibodies (ADAs) | Days 1 through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR